CLINICAL TRIAL: NCT06139406
Title: A Phase 1, First-in-human Study of JNJ-87801493 in Combination With CD3 T-Cell Engagers in Participants With Relapsed/Refractory B-cell Non-Hodgkin Lymphoid Malignancies (NHLs)
Brief Title: A Study of JNJ-87801493 in Combination With T-Cell Engagers in Participants With B-cell Non-Hodgkin Lymphoid (NHLs) Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 87801493LYM1001; 87801493LYM1001 (Other: Janssen Research & Development, LLC); 2023-505165-93-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1: Dose escalation (Experimental): Participants will receive one cycle of TCE monotherapy (step up dosing) with either JNJ-80948543 or JNJ-75348780 followed by initiation of combination therapy with JNJ-87801493 at least one week later.
  Interventions: Drug: JNJ-87801493; Drug: JNJ-80948543; Drug: JNJ-75348780
- Part 2:Dose expansion (Experimental): Participants with specific B-cell NHL histologies will receive recommended phase 2 regimen (RP2R) of JNJ-87801493 with TCE as determined in Part 1.
  Interventions: Drug: JNJ-87801493; Drug: JNJ-80948543; Drug: JNJ-75348780

INTERVENTIONS:
Drug: JNJ-87801493 — JNJ-87801493 will be administered subcutaneously.
Drug: JNJ-80948543 — JNJ-80948543 will be administered subcutaneously.
Drug: JNJ-75348780 — JNJ-75348780 will be administered subcutaneously.

SUMMARY:
The purpose of this study is to characterize safety and to determine the recommended phase 2 regimen (RP2R) for JNJ-87801493 in combination with T-cell engagers (TCEs) [Part A: Dose Escalation] and to further assess the safety of JNJ-87801493 at the RP2R in combination with TCEs [Part B: Dose Expansion].

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of B-cell NHL. All participants in part 1 must have relapsed or refractory disease with no other approved therapies available that would be more appropriate in the investigator's judgment. In Part 2, participants with diffuse large B-cell lymphoma (DLBCL) or other high-grade B cell lymphoma and participants with transformed lymphoma from low-grade B cell malignancies who relapsed or failed to respond to only one prior systemic treatment regimen can be included
* Part 1 participants must have evaluable or measurable disease and Part 2 participants must have measurable disease; all as defined by the Lugano criteria for non-Hodgkin lymphoid malignancies (NHL) and the international workshop on Waldenstrom's Macroglobulinemia (IWWM-6) for WM
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Hematologic laboratory parameters must meet the required criterias and the values must be without a transfusion or growth factors for at least 7 days prior to the first dose of study drug
* Participants of childbearing potential must have a negative highly sensitive serum pregnancy test (beta (β)-human chorionic gonadotropin) at screening and within 72 hours of the first dose of study treatment and must agree to further serum or urine pregnancy tests during the study.

Exclusion Criteria:

* Known active central nervous system involvement (CNS) or leptomeningeal involvement. CNS involvement may be allowed in specific cohorts as determined by the Study Evaluation Team (SET)
* Prior solid-organ transplantation
* Prior treatment with JNJ-80948543 and/or JNJ-75348780. In addition, history of known allergies, hypersensitivity, or intolerance to either JNJ-80948543, JNJ-75348780, or JNJ-87801493 or its excipients
* Chemotherapy, targeted therapy, or immunotherapy within 2 weeks before the first dose of study treatment. For investigational agents where the half-life is known, there should be a treatment-free window of at least 2 weeks or 5 half-lives. For checkpoint blockade therapy (example, anti-programmed cell death protein-1 [anti-PD-1]), a washout period of up to 6 weeks may be considered
* Malignancy diagnosis other than the disease under study within 1 year prior to screening. Exceptions are squamous and basal cell carcinoma of the skin, carcinoma in situ of the cervix and any malignancy that is considered cured or has minimal risk of recurrence within 1 year of first dose of the study drugs in the opinion of both the investigator and sponsor's medical monitor
* Autoimmune or inflammatory disease requiring systemic corticosteroids or other immunosuppressive agents within 1 year prior to first dose of study treatment
* Evidence of active viral, bacterial, or uncontrolled systemic fungal infection requiring systemic treatment within 7 days before the first dose of study treatment
* Abnormal cardiac function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose Limiting Toxicity (DLTs) | Up to 2 years 7 months
  Number of participants with DLTs will be reported. The DLTs are drug-related toxicities and are defined as any of the following: fatal toxicity, high grade non-hematologic toxicity, or hematologic toxicity
Part 1 and 2: Percentage of Participants with Adverse Events (AEs) by Severity | Up to 2 years 7 months
  An AE is any untoward medical occurrence in a clinical study participant administered an investigational or non-investigational product and it does not necessarily have a causal relationship with the investigational product. Severity for AEs will be specified as per: NCI-CTCAE grades which are Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (potentially life-threatening) and; American Society for Transplantation and Cellular Therapy (ASTCT) guidelines which is Grade 5 (death related to adverse event); Cytokine release syndrome (CRS) and associated neurologic toxicity events (immune effector cell-associated neurotoxicity syndrome events [ICANS]).

SECONDARY OUTCOMES:
Serum Concentration for JNJ-87801493, JNJ-80948543 and JNJ-75348780 | Up to 2 years 7 months
  Serum Concentration for JNJ-87801493, JNJ-80948543 and JNJ-75348780 will be reported.
Area Under the Curve (AUCtau) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 | Up to 2 years 7 months
  AUC tau is defined as area under the serum concentration-time curve during a dosing interval (tau).Area under the serum concentration curve (AUCtau) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 will be reported.
Maximum Serum Concentration (Cmax) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 | Up to 2 years 7 months
  Maximum observed serum concentration (Cmax) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 will be reported.
Minimum Serum Concentration (Cmin) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 | Up to 2 years 7 months
  Minimum observed serum concentration (Cmin) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 will be reported.
Area Under the Curve (AUC[0-t]) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 | Up to 2 years 7 months
  Area under the curve from time zero to t (AUC[0-t]) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 will be reported.
Half-life (t1/2) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 | Up to 2 years 7 months
  Half-life (t1/2) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 will be reported.
Time to Reach Cmax (Tmax) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 | Up to 2 years 7 months
  Tmax is the time to reach maximum observed serum concentartion for JNJ-87801493, JNJ-80948543 and JNJ-75348780.
Apparent Total Body Clearance (CL/F) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 | Up to 2 years 7 months
  Apparent total body clearance (CL/F) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 will be reported.
Apparent Volume of Distribution (V/F) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 | Up to 2 years 7 months
  Apparent volume of distribution (V/F) for JNJ-87801493, JNJ-80948543 and JNJ-75348780 will be reported.
Number of Participants with Presence of Anti-JNJ-87801493, Anti-JNJ- 80948543 and Anti-JNJ-75348780 Antibodies | Up to 2 years 7 months
  Number of participants with presence of antibodies binding to JNJ-87801493 or each combination partner (JNJ- 80948543 and JNJ-75348780).
Overall Response as Assessed by the Investigator | Up to 2 years 7 months
  Overall response is defined as a best response of partial response (PR) or better.
Complete Response (CR) as Assessed by the Investigator | Up to 2 years 7 months
  Complete response (CR) is defined as a best response of CR.
Very Good Partial Response (VGPR) or better for Waldenström Macroglobulinemia (WM) Participants as Assessed by the Investigator | Up to 2 years 7 months
  Very good partial response (VGPR) or better is defined as a best response of VGPR or better.
Time to Response (TTR) as Assessed by the Investigator | Up to 2 years 7 months
  Time to response (TTR) is defined for participants who achieve a response of PR or better as the time from the first dose of any study drug to the first response of PR or better.
Duration of Response (DOR) as Assessed by the Investigator | Up to 2 years 7 months
  Duration of response (DOR) is defined for participants who achieved a response of PR or better as the time from the first efficacy evaluation at which the participant meet all criteria for a response of PR or better to the date of first documented evidence of progressive disease or death.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (12):
- Australia (4):
  - Austin Hospital, Heidelberg
  - The Alfred Hospital, Melbourne
  - Linear Clinical Research Ltd, Nedlands
  - Scientia Clinical Research, Randwick
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Sourasky (Ichilov) Medical Center, Tel Aviv
- Spain (4):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency